CLINICAL TRIAL: NCT03273153
Title: A Phase III, Open-Label, Multicenter, Two Arm, Randomized Study to Investigate the Efficacy and Safety of Cobimetinib Plus Atezolizumab Versus Pembrolizumab in Patients With Previously Untreated Advanced BRAF V600 Wild-Type Melanoma
Brief Title: A Study of Cobimetinib Plus Atezolizumab Versus Pembrolizumab in Participants With Previously Untreated Advanced BRAFv600 Wild-Type Melanoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to benefit/risk analysis.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO39722; 2016-004387-18 (EudraCT Number)
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Advanced BRAFV600 Wild-type Melanoma
MeSH Terms: interventions — cobimetinib; atezolizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cobimetinib and Atezolizumab (Experimental): Participants will receive 60 mg of cobimetinib orally from Days 1 to 21 along with 840 mg of atezolizumab by intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle until investigator-determined disease progression, unacceptable toxicity, death, patient or physician decision to withdraw, or pregnancy, whichever occurs first. There will be no cobimetinib administration for 7 days (Days 22-28) in each cycle.
  Interventions: Drug: Cobimetinib; Drug: Atezolizumab
- Pembrolizumab (Active Comparator): Participants will receive 200 mg of pembrolizumab administered by IV infusion every 3 weeks (Q3W) until investigator-determined disease progression, unacceptable toxicity, death, patient or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib 60 mg tablets orally once daily on a 21 days on, 7 days off schedule.
  Arms: Cobimetinib and Atezolizumab
Drug: Atezolizumab — Atezolizumab 840 mg as IV infusion once in every 2 weeks.
  Arms: Cobimetinib and Atezolizumab
Drug: Pembrolizumab — Pembrolizumab 200 mg as IV infusion once in every 3 weeks.
  Arms: Pembrolizumab

SUMMARY:
This is a Phase III, multicenter, open-label, randomized study designed to evaluate the efficacy, safety, and pharmacokinetics of cobimetinib plus atezolizumab compared with pembrolizumab in treatment-naive participants with advanced BRAFV600 wild-type melanoma.

ELIGIBILITY:
Inclusion Criteria:

Disease-Specific Inclusion Criteria

* Histologically confirmed locally advanced and unresectable or metastatic melanoma
* Naive to prior systemic anti-cancer therapy for melanoma
* Documentation of BRAFV600 wild-type status in melanoma tumor tissue through use of a clinical mutation test approved by the local health authority
* A representative, formalin-fixed, paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or 20 slides containing unstained, freshly cut, serial sections must be submitted along with an associated pathology report prior to study entry. If 20 slides are not available or the tissue block is not of sufficient size, the patient may still be eligible for the study, after discussion with and approval by the Medical Monitor
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Age >=18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Histologically or cytologically confirmed BRAFV600 wild-type melanoma
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy >=3 months
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent or use at least two forms of effective contraceptive with a failure rate of < 1% per year during the treatment period and for at least 3 months after the last dose of cobimetinib and at least 5 months after the last dose of atezolizumab or pembrolizumab
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures (e.g. condom), and agreement to refrain from donating sperm, for at least 3 months after the last dose of cobimetinib
* Willingness and ability of patients to report selected study outcomes (e.g., GHS and HRQoL) using an electronic device or paper backup questionnaires.

Exclusion Criteria:

General Exclusion Criteria

* Inability to swallow medications
* Malabsorption condition that would alter the absorption of orally administered medications
* Pregnancy, breastfeeding, or intention of becoming pregnant during the study
* History of severe hypersensitivity reactions to components of the cobimetinib, atezolizumab, or pembrolizumab formulations
* Current or recent treatment with therapeutic antibiotics, live attenuated vaccines or systemic immunostimulatory/immunosuppresive medication
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study Cancer-Related Exclusion Criteria
* Ocular melanoma
* Major surgery or radiotherapy within 21 days prior to Day 1 of Cycle 1 or anticipation of needing such procedure while receiving study treatment
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage more than once every 28 days
* Active or untreated central nervous system (CNS) metastases Exclusions Related to Cardiovascular Disease
* Unstable angina, new-onset angina within last 3 months, myocardial infarction within the last 6 months prior to Day 1 of Cycle 1, or current congestive heart failure classified as New York Heart Association Class II or higher
* Left ventricular ejection fraction (LVEF) below institutional lower limit of normal or <50%, whichever is lower
* Poorly controlled hypertension, defined as sustained, uncontrolled, non-episodic baseline hypertension consistently above 159/99 mmHg despite optimal medical management
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third degree heart block, or evidence of prior myocardial infarction Exclusions Related to Infections
* HIV infection
* Active tuberculosis infection
* Severe infections within 4 weeks prior to Day 1 of Cycle 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of clinically relevant infection within 2 weeks prior to Day 1 of Cycle 1
* Treatment with oral or IV antibiotics within 2 weeks prior to Day 1 of Cycle 1
* Active or chronic viral hepatitis B or C infection Exclusions Related to Ocular Disease
* Known risk factors for ocular toxicity Exclusions Related to Autoimmune Conditions and Immunomodulatory Drugs
* Active or history of autoimmune disease or immune deficiency
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Treatment with systemic immunosuppressive medications within 2 weeks prior to Day 1, Cycle 1 Exclusions Related to Other Medical Conditions or Medications
* Active malignancy (other than melanoma) or a prior malignancy within the past 3 years
* Any Grade >=3 hemorrhage or bleeding event within 28 days of Day 1 of Cycle 1
* History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months prior to Day 1
* Proteinuria >3.5 gm/24 hr
* Consumption of foods, supplements, or drugs that are strong or moderate CYP3A4 enzyme inducers or inhibitors at least 7 days prior to Day 1 of Cycle 1 and during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (121):
- United States (23):
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC Norris Cancer Center, Los Angeles, California
  - USC Norris Cancer Center; USC Oncology Hematology Newport Beach, Newport Beach, California
  - University of California at Irvine Medical Center; Department of Oncology, Orange, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital;Hematology/ Oncology, Boston, Massachusetts
  - University of Michigan; Michigan Institute for Clinical and Health Research (MICHR), Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center; Hematology/Oncology, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Forsythe Memorial Hospital Inc., dba Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - TriHealth Hatton Institute; Surgical Education, Cincinnati, Ohio
  - St. Luke's University Health network, Bethlehem, Pennsylvania
  - Thomas Jefferson University Hospital;Medical Oncology, Philadelphia, Pennsylvania
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - M.D Anderson Cancer Center; Uni of Texas At Houston, Houston, Texas
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
- Australia (5):
  - Cairns Base Hospital, Cairns, Queensland
  - Townsville General Hospital, Douglas, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (2):
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
- France (16):
  - Hopital Avicenne; Dermatologie, Bobigny
  - Hopital Saint Andre CHU De Bordeaux; Dermatologie, Bordeaux
  - Chu Site Du Bocage;Dermatologie, Dijon
  - CHU de Grenoble - Hôpital Nord, Grenoble
  - Centre Hospitalier Le Mans; Dermatologie, Le Mans
  - Hopital Claude Huriez; Sce Dermatologie, Lille
  - Hopital Timone Adultes; Dermatologie, Marseille
  - CHU de Nantes; Cancéro-dermatologie, Nantes
  - Hopital l Archet 2; Ginestriere, Service de; Dermatologie, Nice
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - Hopital Saint Louis; Dermatologie 1, Paris
  - Hopital Robert Debre; DERMATOLOGIE, Reims
  - Centre Eugene Marquis; Service d'oncologie, Rennes
  - Hopital Charles Nicolle; Dermatologie Serv., Rouen
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse
  - Institut Gustave Roussy; Dermatologie, Villejuif
- Germany (13):
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Dermatologie, Dresden
  - HELIOS Klinikum Erfurt; Klinik für Dermatologie & Allergologie, Erfurt
  - Universitatsklinikum Essen; Klinik für Dermatologie, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - SRH Wald-Klinikum Gera; Klinik für Hautkrankheiten und Allergologie, Gera
  - Medizinische Hochschule Hannover; Klinik für Dermatologie, Allergologie und Venerologie, Hanover
  - UKSH Kiel; Klinik für Dermatologie, Venerologie und Allergologie, Kiel
  - Universitatsklinikum Mainz; Klinik und Poliklinik fur Dermatologie, Mainz
  - Klinikum Mannheim Klinik fuer Dermatologie, Venerologie und Allergologie, Mannheim
  - Johannes Wesling Klinikum Minden; Hämatologie, Onkologie, Hämostaseologie und Palliativmedizin, Minden
  - Klinikum der Ludwigs-Maximilians-Universität München; Dermatologie, München
  - Fachklinik Hornheide; Dermatologie, Münster
  - Zentrum für Dermatoonkologie, Universitäts-Hautklinik Tübingen, Tübingen
- Greece (4):
  - Anticancer Hospital Ag. Savas ; 2Nd Dept. of Oncology - Internal Medicine, Athens
  - Laiko General Hospital Athen, Athens
  - Metropolitan Hospital; Dept. of Oncology, Pireaus
  - Bioclinic Thessaloniki, Thessaloniki
- Hungary (3):
  - Orszagos Onkologiai Intezet; Borgyogyaszati Osztaly, Budapest
  - Pecsi Tudomanyegyetem AOK; Borgyogyaszati Klinika, Pécs
  - University of Szeged Szent-Györgyi Albert Clinical Center; Department of Dermatology and Allergology, Szeged
- Italy (11):
  - A.O.U. Cons. Policlinico Bari - Consorzlale Policlinico; Scienze Biomediche e Oncologia Umana, Bari, Apulia
  - Azienda Osp Uni Seconda Università Degli Studi Di Napoli; Unità Operativa Oncologia Medica, Napoli, Campania
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale; Oncologia Medica B, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - IFO - Istituto Regina Elena; Oncologia Medica, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Azienda Ospedaliero - Universitaria Pisana U.O. Oncologia Medica 2 Universitaria - Polo Oncologico, Pisa, Tuscany
  - IOV - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- Netherlands (4):
  - Antoni Van Leeuwenhoek Ziekenhuis; Inwendige Geneeskunde, Amsterdam
  - Amphia Ziekenhuis, locatie Langendijk;Oncology, Breda
  - Erasmus Mc - Daniel Den Hoed Kliniek; Interne Oncologie, Rotterdam
  - Zuyderland ziekenhuis locatie Geleen, Sittard-Geleen
- Poland (6):
  - Copernicus Podmiot Medyczny Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu., Poznan
  - Zachodniopomorskie Centrum Onkologii, Osrodek Innowacyjnosci, Rozwoju i Badan Klinicznych, Szczecin
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
  - Dolnośląskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw
- Russia (4):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - St. Petersburg Oncology Hospital, Saint Petersburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (15):
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Clinica Universitaria de Navarra; Servicio de oncología, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Oncología, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- United Kingdom (8):
  - BRISTOL ONCOLOGY CENTRE; CLINICAL TRIALS UNIT; R & D department, Bristol
  - Western General Hospital; Edinburgh Cancer Center, Edinburgh
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - University College London Hospital, London
  - Guys & St Thomas Hospital; Department of Oncology, London
  - University Hospitals of North Midlands NHS Trust-Royal Stoke University Hospital, Stoke-on-Trent
  - Singleton Hospital; Pharmacy, Swansea
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] de Azevedo SJ, de Melo AC, Roberts L, Caro I, Xue C, Wainstein A. First-line atezolizumab monotherapy in patients with advanced BRAFV600 wild-type melanoma. Pigment Cell Melanoma Res. 2021 Sep;34(5):973-977. doi: 10.1111/pcmr.12960. Epub 2021 Feb 15. PMID 33476492

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Participants received 200 mg of intravenous (IV) pembrolizumab every 3 weeks (Q3W) until investigator-determined disease progression, unacceptable toxicity, death, patient or physician decision to withdraw, or pregnancy, whichever occurred first.
- Cobimetinib and Atezolizumab: Participants received 60 mg of cobimetinib by mouth (PO) on a 21 days on, 7 days off schedule (dosing on Days 1-21, followed by no dosing on Days 22-28) plus 840 mg of atezolizumab by IV infusion of Days 1 and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Started | 224 | 222
Completed | 0 | 0
Not Completed | 224 | 222
Not completed — Adverse Event | 1 | 2
Not completed — Missing | 0 | 2
Not completed — Other | 3 | 2
Not completed — Symptomatic Deterioration | 0 | 1
Not completed — Progressive Disease | 6 | 5
Not completed — Physician Decision | 1 | 3
Not completed — Study Terminated by Sponsor | 112 | 102
Not completed — Withdrawal by Subject | 26 | 25
Not completed — Protocol Deviation | 3 | 0
Not completed — Lost to Follow-up | 6 | 11
Not completed — Death | 66 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab | Total
Number analyzed (Participants) | 224 | 222 | 446
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (12.9) | 63.6 (13.1) | 63.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 93 | 176
  Male | 141 | 129 | 270
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 15 | 22
  Not Hispanic or Latino | 190 | 180 | 370
  Unknown or Not Reported | 27 | 27 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 198 | 188 | 386
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Determined by the Independent Review Committee (IRC)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression, as determined by an IRC according to RECIST v1.1, or death from any cause, whichever occurs first. Progressive disease (PD) for target lesion: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/=5 mm. PD for non-target lesion: Unequivocal progression of existing non-target lesions.
Time Frame: Every 8 weeks (wks) from Day (D) 1 of Cycle (C) 1 through approximately 16 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 224 | 222
Months | 5.7 [3.7 to 9.6] | 5.5 [3.8 to 7.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Cobimetinib and Atezolizumab; Test type: Superiority; p = 0.2954, Regression, Cox; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.88 to 1.50]

2. Secondary Outcome: PFS as Determined by the Investigator
Description: PFS is defined as the time from randomization to the first occurrence of disease progression, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. Progressive disease (PD) for target lesion: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/=5 mm. PD for non-target lesion: Unequivocal progression of existing non-target lesions.
Time Frame: Every 8 weeks (wks) from Day (D) 1 of Cycle (C) 1 through approximately 16 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 224 | 222
Months | 7.2 [3.8 to 10.1] | 5.6 [3.9 to 6.6]

3. Secondary Outcome: Objective Response as Determined by the Investigator
Description: Objective response rate is defined as the percentage of participants with a complete response (CR) or a partial response (PR) on two consecutive occasions >/=4 weeks apart, as determined by the investigator through the use of RECIST v1.1. For target lesion, CR: the disappearance of all target lesions, any pathological lymph nodes must have a reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. For non-target lesion, CR: the disappearance of all non-target lesions and (if applicable) normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis).
Time Frame: Every 8 weeks (wks) from Day (D) 1 of Cycle (C) 1 through approximately 16 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 221 | 222
Percentage of Participants | 36.7 [30.29 to 43.38] | 27.9 [22.13 to 34.32]

4. Secondary Outcome: Objective Response as Determined by IRC
Description: Objective response, defined as a complete response or partial response on two consecutive occasions ≥4 weeks apart, as determined by IRC according to RECIST v1.1
Time Frame: Every 8 weeks (wks) from Day (D) 1 of Cycle (C) 1 through approximately 16 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 206 | 204
Percentage of Participants | 31.6 [25.27 to 38.38] | 26.0 [20.11 to 32.57]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the proportion of participants with a complete response, a partial response, or stable disease at 16 weeks. For target lesion, CR: the disappearance of all target lesions, any pathological lymph nodes must have a reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. For non-target lesion, CR: the disappearance of all non-target lesions and (if applicable) normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis). Stable disease (SD): neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD.
Time Frame: Week 16
Population: The analysis for this outcome measure was limited to participants meeting the criteria provided in the description.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 221 | 222
Percentage of Participants
  Investigator-assessed | 49.8 [43.00 to 56.56] | 46.8 [40.14 to 53.64]
  IRC-assessed: number analyzed (Participants) | 206 | 204
  IRC-assessed | 44.2 [37.28 to 51.24] | 45.6 [38.62 to 52.69]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: From randomization up to approximately 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 224 | 222
Months | 29.3 [21.5 to NA] — Values are not estimable due to an insufficient number of participants with the event. | NA [24.1 to NA] — Values are not estimable due to an insufficient number of participants with the event.

7. Secondary Outcome: Duration of Objective Response Determined by the IRC
Description: Duration of objective response, defined as the time from the first occurrence of a documented objective response to disease progression, as determined by an IRC according to RECIST v1.1, or death from any cause, whichever occurs first.
Time Frame: Every 8 weeks (wks) from Day (D) 1 of Cycle (C) 1 through approximately 16 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 206 | 204
Months | NA [NA to NA] — Values are not estimable due to an insufficient number of participants with the event. | NA [9.2 to NA] — Values are not estimable due to an insufficient number of participants with the event.

8. Secondary Outcome: Duration of Objective Response Determined by the Investigator
Description: Duration of objective response is defined as the time from the first occurrence of a documented objective response to disease progression, as determined by the investigator through use of RECIST v1.1, or death from any cause, whichever occurs first.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 221 | 222
Months | NA [NA to NA] — Values are not estimable due to an insufficient number of participants with the event. | NA [9.2 to NA] — Values are not estimable due to an insufficient number of participants with the event.

9. Secondary Outcome: Two-year Landmark Survival
Description: Two-year landmark survival is defined as the rate of survival at 2 years. Two-year landmark survival is defined as the rate of survival at 2 years and was calculated using Kaplan-Meier analysis, which is commonly used to estimate the probability of an event at time 't.'
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 224 | 222
Percentage | 57.88 [48.25 to 67.52] | 60.19 [51.58 to 68.79]

10. Secondary Outcome: Change From Baseline in Health-related Quality of Life (HRQoL) Scores
Description: HRQoL scores are assessed through global health status (GHS)/ quality of life (QoL) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C30). These are based on questions 29 and 30 of the EORTC QLQ-C30. These questions on global health status/QoL scale are coded on 7-point scale (1=very poor to 7=excellent). Raw scores will be linearly transformed to obtain the score ranging from 0 to 100, where higher score represents a higher ("better") level of functioning.
Time Frame: Up to approximately 16 months. Follow up is reported at weeks after participant treatment discontinuation, which could occur at any time during the study. Total time frame does not exceed 16 months.
Population: The analysis population for this endpoint was the patient reported outcome (PRO) population evaluable participants for EORTC QLQ-C30.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 174 | 160
Units on a Scale
  Baseline value: number analyzed (Participants) | 173 | 160
  Baseline value | 73.27 (20.41) | 73.85 (19.73)
  Week 4: number analyzed (Participants) | 131 | 124
  Week 4 | -2.99 (17.05) | -9.14 (20.83)
  Week 8: number analyzed (Participants) | 119 | 104
  Week 8 | -3.15 (18.67) | -5.21 (18.18)
  Week 12: number analyzed (Participants) | 94 | 97
  Week 12 | -1.77 (19.93) | -7.65 (21.20)
  Week 16: number analyzed (Participants) | 79 | 75
  Week 16 | 1.16 (15.02) | -6.44 (20.58)
  Week 20: number analyzed (Participants) | 74 | 66
  Week 20 | 1.69 (17.50) | -6.31 (19.17)
  Week 24: number analyzed (Participants) | 59 | 57
  Week 24 | -1.84 (19.82) | -2.49 (15.98)
  Week 28: number analyzed (Participants) | 44 | 41
  Week 28 | 2.46 (19.07) | -3.86 (19.10)
  Week 32: number analyzed (Participants) | 38 | 34
  Week 32 | -0.88 (22.41) | -4.66 (20.94)
  Week 36: number analyzed (Participants) | 24 | 25
  Week 36 | 4.17 (20.56) | -6.00 (18.24)
  Week 40: number analyzed (Participants) | 15 | 18
  Week 40 | 7.22 (19.38) | -4.63 (21.62)
  Week 44: number analyzed (Participants) | 18 | 10
  Week 44 | 0.46 (19.27) | 1.67 (12.91)
  Week 48: number analyzed (Participants) | 12 | 7
  Week 48 | 7.64 (13.04) | 0.00 (15.96)
  Week 52: number analyzed (Participants) | 5 | 4
  Week 52 | 1.67 (12.36) | 8.33 (15.21)
  Week 56: number analyzed (Participants) | 6 | 4
  Week 56 | -11.11 (17.21) | -2.08 (4.17)
  Week 60: number analyzed (Participants) | 2 | 2
  Week 60 | -8.33 (11.79) | -4.17 (5.89)
  Week 64: number analyzed (Participants) | 1 | 0
  Week 64 | 33.33 (NA) — Value is NA due to an insufficient number of participants with the event at this timepoint. |
  Treatment Discontinuation: number analyzed (Participants) | 95 | 78
  Treatment Discontinuation | -6.05 (22.53) | -14.42 (25.68)
  Follow-up 4: number analyzed (Participants) | 12 | 11
  Follow-up 4 | -7.64 (14.85) | -2.27 (18.67)
  Follow-up 8: number analyzed (Participants) | 31 | 13
  Follow-up 8 | -14.25 (21.96) | -14.10 (24.15)
  Follow-up 12: number analyzed (Participants) | 23 | 12
  Follow-up 12 | -21.38 (24.34) | -24.31 (28.08)
  Follow-up 16: number analyzed (Participants) | 17 | 12
  Follow-up 16 | -13.73 (19.53) | -23.61 (23.26)
  Follow-up 20: number analyzed (Participants) | 16 | 6
  Follow-up 20 | -20.83 (26.53) | -8.33 (12.91)
  Follow-up 24: number analyzed (Participants) | 8 | 5
  Follow-up 24 | -17.71 (29.36) | -10.00 (14.91)
  Follow-up 28: number analyzed (Participants) | 6 | 2
  Follow-up 28 | -27.78 (22.15) | -16.67 (23.57)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to approximately 16 months
Measure: Number; unit: Number of Participants
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 216 | 220
Number of Participants | 195 | 218

12. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital signs will include temperature, pulse rate, respiratory rate, and systolic and diastolic blood pressure.
Time Frame: From baseline up to approximately 3 years
Population: N for each assessment = participants without abnormalities at baseline or with missing baseline values
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 216 | 220
Participants
  Sitting diastolic blood pressure - low: number analyzed (Participants) | 210 | 214
  Sitting diastolic blood pressure - low | 41 | 42
  Sitting diastolic blood pressure - high: number analyzed (Participants) | 150 | 138
  Sitting diastolic blood pressure - high | 77 | 85
  Sitting systolic blood pressure - low | 4 | 7
  Sitting systolic blood pressure - high: number analyzed (Participants) | 69 | 60
  Sitting systolic blood pressure - high | 53 | 47
  Pulse rate - low: number analyzed (Participants) | 199 | 196
  Pulse rate - low | 58 | 67
  Pulse rate - high: number analyzed (Participants) | 208 | 214
  Pulse rate - high | 13 | 27
  Respiratory rate - low: number analyzed (Participants) | 209 | 219
  Respiratory rate - low | 8 | 11
  Respiratory rate - high: number analyzed (Participants) | 194 | 200
  Respiratory rate - high | 55 | 52
  Temperature - low: number analyzed (Participants) | 121 | 117
  Temperature - low | 91 | 93
  Temperature - high: number analyzed (Participants) | 213 | 214
  Temperature - high | 20 | 47

13. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Participants with laboratory abnormalities (values outside of a defined range) will be reported.
Time Frame: Up to approximately 16 months
Population: Participants with at least one post-baseline assessment for a given laboratory value were included in this assessment.
Measure: Number; unit: Number of Participants
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 216 | 220
Number of Participants
  SGPT/ALT | 1 | 1
  Amylase: number analyzed (Participants) | 201 | 204
  Amylase | 4 | 5
  SGOT/AST: number analyzed (Participants) | 215 | 220
  SGOT/AST | 0 | 2
  Calcium | 0 | 1
  Creatine Kinase: number analyzed (Participants) | 215 | 220
  Creatine Kinase | 1 | 17
  Creatinine | 1 | 4
  Glucose: number analyzed (Participants) | 210 | 218
  Glucose | 8 | 13
  Triacylglycerol Lipase: number analyzed (Participants) | 197 | 200
  Triacylglycerol Lipase | 8 | 10
  Magnesium: number analyzed (Participants) | 215 | 217
  Magnesium | 3 | 2
  Phosphorus: number analyzed (Participants) | 216 | 217
  Phosphorus | 6 | 10
  Potassium | 1 | 6
  Sodium | 2 | 4
  Uric Acid: number analyzed (Participants) | 179 | 188
  Uric Acid | 36 | 30
  Hemoglobin | 2 | 2
  Lymphocytes Abs: number analyzed (Participants) | 173 | 178
  Lymphocytes Abs | 6 | 15
  Neutrophils, Total, Abs: number analyzed (Participants) | 174 | 179
  Neutrophils, Total, Abs | 0 | 1
  Total Leukocyte Count | 3 | 0

14. Secondary Outcome: Plasma Concentration of Cobimetinib
Time Frame: Days 1 and 15 of Cycle 1
Population: PK data was not available from all participants at all time points due to study continuation or missed PK sampling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/mL
Arm/Group | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 202
nanograms/mL
  Cycle 1 Day 1 | 49.2 (614.7)
  Cycle 1 Day 15 pre-dose: number analyzed (Participants) | 142
  Cycle 1 Day 15 pre-dose | 126 (284.1)
  Cycle 1 Day 15 post-dose: number analyzed (Participants) | 130
  Cycle 1 Day 15 post-dose | 231 (213.3)

15. Secondary Outcome: Serum Concentration of Atezolizumab
Time Frame: Day 1 of Cycles 1, 2, and 3
Population: PK data was not available from all participants at all time points due to study continuation or missed PK sampling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/mL
Arm/Group | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 196
micrograms/mL
  Cycle 1 Day 1 | 256 (35.3)
  Cycle 2 Day 1: number analyzed (Participants) | 163
  Cycle 2 Day 1 | 72.2 (177.1)
  Cycle 3 Day 1: number analyzed (Participants) | 142
  Cycle 3 Day 1 | 126 (104.3)

16. Secondary Outcome: Percentage of Participants With Anti-drug Antibodies (ADAs)
Description: Participants with ADAs during the study relative to the prevalence of ADAs at baseline will be reported.
Time Frame: Day 1 of Cycle 1, 2, 3 and 30 days after treatment discontinuation
Population: Only participants from the Cobimetinib and Atezolizumab arm are included in this endpoint as it is meant to evaluate the immune response to atezolizumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Cobimetinib and Atezolizumab
Number analyzed (Participants) | 210
Percentage of participants | 23.2

ADVERSE EVENTS:
Time Frame: For up to 135 days after the last dose of study drug, or until a new systemic anti-cancer therapy was initiated, whichever occurred first (a maximum of approximately 3 years).
Description: Adverse events (serious and other) were evaluated for the safety-evaluable population, which consisted of all participants who received at least one dose of study treatment. All-cause mortality is reported for the entire study population.
Arm/Group | Pembrolizumab | Cobimetinib and Atezolizumab
All-Cause Mortality (participants affected / at risk) | 68/224 | 70/222
Serious Adverse Events (participants affected / at risk) | 56/216 | 105/220
Other Adverse Events (participants affected / at risk) | 173/216 | 209/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=216) | Cobimetinib and Atezolizumab (N=220)
Diarrhoea (Gastrointestinal disorders) | 2 | 9
Vomiting (Gastrointestinal disorders) | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 12
Asthenia (General disorders) | 3 | 4
Fatigue (General disorders) | 0 | 3
General physical health deterioration (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 3
Diarrhoea infectious (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 3
Seizure (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 2
Autoimmune encephalopathy (Nervous system disorders) | 0 | 1
Encephalitis autoimmune (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Hypotension (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Chorioretinopathy (Eye disorders) | 0 | 2
Visual impairment (Eye disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Immune-mediated neuropathy (Nervous system disorders) | 0 | 1
Autoimmune nephritis (Renal and urinary disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 6
Pneumonia (Infections and infestations) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Chest pain (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypotensive crisis (Vascular disorders) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spleen tuberculosis (Infections and infestations) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Superinfection viral (Infections and infestations) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1
Tonsilitis (Infections and infestations) | 0 | 1
Toxic shock syndrome (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=216) | Cobimetinib and Atezolizumab (N=220)
Anaemia (Blood and lymphatic system disorders) | 17 (18) | 32 (50)
Hyperthyroidism (Endocrine disorders) | 21 (22) | 10 (10)
Hypothyroidism (Endocrine disorders) | 17 (17) | 15 (17)
Abdominal pain (Gastrointestinal disorders) | 18 (22) | 24 (29)
Constipation (Gastrointestinal disorders) | 20 (26) | 32 (36)
Diarrhoea (Gastrointestinal disorders) | 42 (58) | 120 (293)
Dry mouth (Gastrointestinal disorders) | 9 (9) | 18 (19)
Nausea (Gastrointestinal disorders) | 28 (32) | 54 (61)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 14 (19)
Vomiting (Gastrointestinal disorders) | 15 (16) | 41 (53)
Asthenia (General disorders) | 42 (49) | 59 (89)
Fatigue (General disorders) | 42 (54) | 43 (64)
Oedema peripheral (General disorders) | 17 (20) | 50 (76)
Pyrexia (General disorders) | 17 (19) | 65 (87)
Folliculitis (Infections and infestations) | 2 (2) | 15 (24)
Rash pustular (Infections and infestations) | 2 (2) | 11 (12)
Urinary tract infection (Infections and infestations) | 4 (4) | 13 (18)
Alanine aminotransferase increased (Investigations) | 18 (19) | 30 (42)
Amylase increased (Investigations) | 9 (10) | 19 (29)
Aspartate aminotransferase increased (Investigations) | 18 (20) | 42 (57)
Blood creatine phosphokinase increased (Investigations) | 13 (16) | 81 (127)
Blood lactate dehydrogenase increased (Investigations) | 5 (5) | 15 (19)
Lipase increased (Investigations) | 15 (18) | 28 (51)
Decreased appetite (Metabolism and nutrition disorders) | 16 (18) | 30 (35)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (13) | 19 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 (48) | 21 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (29) | 12 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 18 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 11 (12)
Dizziness (Nervous system disorders) | 8 (11) | 18 (23)
Headache (Nervous system disorders) | 17 (19) | 30 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 21 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 18 (24)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 50 (68)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (15) | 15 (21)
Erythema (Skin and subcutaneous tissue disorders) | 9 (12) | 16 (20)
Pruritis (Skin and subcutaneous tissue disorders) | 35 (42) | 44 (64)
Rash (Skin and subcutaneous tissue disorders) | 27 (37) | 90 (154)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7) | 26 (39)
Hypertension (Vascular disorders) | 15 (21) | 24 (29)
Nasopharyngitis (Infections and infestations) | 10 (15) | 12 (13)
Paronychia (Infections and infestations) | 1 (1) | 13 (14)
Weight decreased (Investigations) | 12 (13) | 11 (13)
Paraesthesia (Nervous system disorders) | 6 (6) | 11 (12)
Vitiligo (Skin and subcutaneous tissue disorders) | 19 (20) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03273153/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT03273153/SAP_000.pdf